CLINICAL TRIAL: NCT06949904
Title: The Role of Melatonin as an Adjuvant Therapy in Childhood Pneumonia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mian Muhammad Hassan Ahmed (Other)
Responsible Party: Sponsor-Investigator, Mian Muhammad Hassan Ahmed, Post Graduate Resident, College of Physicians and Surgeons Pakistan
Organization: College of Physicians and Surgeons Pakistan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: F.1-1/2015/ERB/SZABMU/1186
Record Dates: First submitted 2025-03-31; First posted 2025-04-29 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Pneumonia Childhood
Keywords: Pneumonia; Childhood pneumonia; Melatonin
MeSH Terms: conditions — Pneumonia | interventions — Melatonin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard Treatment (No Intervention): Standard treatment - Antibiotic such as ampicillin in a dose of 50mg//kg/dose x TDS
- Adjuvant Therapy (Experimental): Standard Treatment along with Melatonin @ 1 mg/dose in infants and 2.5 to 3mg/dose in children three times a day for 14 days
  Interventions: Drug: Melatonin

INTERVENTIONS:
Drug: Melatonin — 1 mg/dose in infants and 2.5 to 3mg/dose in children three times a day for 14 days
  Arms: Adjuvant Therapy

SUMMARY:
The goal of this study is to compare the mean length of hospital stay between children with pneumonia receiving melatonin as an adjuvant therapy and those receiving standard of care alone.

The hypothesis is that combining oral melatonin with standard treatment can reduce the length of hospital stay as compared to standard of care alone.

The control group will receive standard treatment (antibiotic) while the intervention group will receive standard treatment plus melatonin for 14 days.

DETAILED DESCRIPTION:
OPERATIONAL DEFINITION:

Pneumonia: defined as patient having fast breathing;

* 50 breaths/min in a child aged 2-11 months
* 40 breaths/min in a child aged 1-5 years Chest in-drawing

Severe Pneumonia: defined as patient having cough or difficulty in breathing with:

Oxygen saturation < 90% or central cyanosis Severe respiratory distress (e.g. grunting, very severe chest in-drawing) Signs of pneumonia with a general danger sign (inability to breastfeed or drink, lethargy or reduced level of consciousness, convulsions) Length of Hospital Stay: measured in days from the day of admission to the day of discharge for both groups.

Discharge Criteria: Discharge criteria for children who have been admitted to the hospital include:

Improvement of vital signs Ability to maintain adequate fluid and nutrition orally Ability to maintain oxygen saturation ≥90 percent in room air Overall clinical improvement including level of activity, appetite, and decreased fever

OPERATIONAL DEFINTION:

Pneumonia: defined as patient having fast breathing;

* 50 breaths/min in a child aged 2-11 months
* 40 breaths/min in a child aged 1-5 years Chest in-drawing

Severe Pneumonia: defined as patient having cough or difficulty in breathing with:

Oxygen saturation < 90% or central cyanosis Severe respiratory distress (e.g. grunting, very severe chest in-drawing) Signs of pneumonia with a general danger sign (inability to breastfeed or drink, lethargy or reduced level of consciousness, convulsions) Length of Hospital Stay: measured in days from the day of admission to the day of discharge for both groups.

Discharge Criteria: Discharge criteria for children who have been admitted to the hospital include:

Improvement of vital signs Ability to maintain adequate fluid and nutrition orally Ability to maintain oxygen saturation ≥90 percent in room air Overall clinical improvement including level of activity, appetite, and decreased fever

RESEARCH METHODOLOGY:

Study design: Randomized Controlled Clinical Trial (RCT) Setting: It will be conducted at Children Hospital, Pakistan Institute of Medical Sciences (PIMS), Islamabad, Pakistan.

Study duration: Approx. 6 months after approval of synopsis. Sample size: Sample size is calculated based on a previous study on the same topic by using WHO sample size calculator; 60 in total having 30 in each group with level of significance 5%, power of test 80%. The median hospital discharge time was 15 days (range: 13-17) for the melatonin group and 21 days (range: 14-24) for the control group (9).

Sampling technique: Consecutive sampling

DATA COLLECTION PROCEDURE:

Prior to the study, healthcare professionals working in emergency departments/outpatient clinics will receive training on their respective roles, responsibilities and study protocols. The clinician will identify eligible patients and provide them with written and verbal information about the study. The parent/legal guardian of the patient will provide informed consent while the patient will provide informed assent if appropriate. After obtaining consent, the patients will be randomized. The control group will receive standard treatment (antibiotic such as ampicillin at a dose of 150mg/kg/day divided every 8 hours), while the intervention group will receive standard treatment plus melatonin for 14 days at the dose of 1 mg/dose in infants and 2.5 to 3mg/dose in children three times a day for 14 days. The patients who will not take more than 10% of the medication will be excluded from the study. The follow-up period will be 2 weeks for all patients.

DATA ANALYSIS PROCEDURE:

Once data collection is complete, the questionnaires will be checked for completeness and consistency by the data collectors. The normality distribution of variables will be evaluated using the Kolmogorov-Smirnov test. Qualitative variables (Gender, socioeconomic status and symptoms (fever, cough, breathing difficulty, decreased oral intake, fits, level of consciousness and persistent vomiting, pneumonia and severe pneumonia)) will be presented as frequencies and percentages (%). Quantitative variables (Age, weight, heart rate, respiratory rate, blood pressure, temperature, oxygen saturation, laboratory parameters (total leukocyte count, hemoglobin, neutrophils, lymphocytes, platelets, C-reactive protein, pH, PCO, P02, HCO3) and length of hospital stay) will be presented as mean ± standard deviation (SD). Both groups (melatonin and non-melatonin) will be compared for length of hospital stay by using independent sample t-test. Effect modifiers like age, gender, socioeconomic status, weight, and pneumonia/ severe pneumonia will be stratified using post stratified independent sample t-test. Statistical analyses will be conducted using SPSS software version 25.0, with a significance level of p-value <0.05.

ELIGIBILITY:
Inclusion Criteria:

* 1 month to 12 years
* Both genders
* Patient diagnosed as having pneumonia or severe pneumonia according to WHO definition

Exclusion Criteria:

* Hospitalized within 14 days prior to the study
* Known TB exposure
* Active varicella or herpes simplex infection
* Allergy to the study medication
* Currently taking melatonin
* Any non pneumonia acute medical illness which requires antibiotic treatment as per local standard of care
* Galactose intolerance, the lapp-lactase deficiency or glucose-galactose malabsorption
* Significant co-morbid disease: lung, cardiac, immune, liver, endocrine, neurological or psychiatric

Ages: 1 Month to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | 14 days
  The primary outcome is the length of hospital stay, measured in days, from admission to discharge. The mean and standard deviation of hospital stay will be calculated for both groups (melatonin and non-melatonin) and compared using an independent sample t-test.

CONTACTS AND LOCATIONS:
Locations (1):
- Pakistan Institute of Medical Sciences, Islamabad, Islamabad, Pakistan

IPD SHARING:
Plan to Share IPD: Yes